CLINICAL TRIAL: NCT07234097
Title: The Influence of Music on perceiVed paIn and leVels of Anxiety whiLe unDergoing transperIneal Prostate Biopsy: the VIVALDI Trial
Acronym: VIVALDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Boeri, Dr, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VIVALDI
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Pain Management
Keywords: pain management; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Group submitted to prostate biopsy with music
  Interventions: Other: Music intervention
- No music (No Intervention): Group submitted to prostate biopsy without music

INTERVENTIONS:
Other: Music intervention — music during the biopsy
  Arms: Music

SUMMARY:
Prostate biopsy is the key examination for the histological diagnosis of prostate cancer. This procedure can be performed via the transrectal (TR) or transperineal (TP) approach. Current Guidelines recommend the transperineal route because it is associated with fewer infectious complications compared to the transrectal approach. However, when the same type of anesthesia is used, the transperineal approach is more painful.

Several strategies have been developed to improve pain management during TR biopsy. Some studies have shown that allowing patients to listen to music during the procedure can reduce perceived pain and stress. However, this effect has never been investigated in TP biopsies, which are now the gold standard and generally more painful than TR biopsies.

Primary Objective:

To evaluate the reduction in pain levels in patients undergoing transperineal prostate biopsy with the aid of music compared to patients undergoing the same procedure without music.

Secondary Objectives:

To evaluate the reduction in stress levels related to the procedure in patients undergoing transperineal prostate biopsy with music compared to those without music.

To evaluate the reduction in the use of painkillers and sedatives during the procedure in patients undergoing transperineal biopsy with music compared to those without.

To assess pain management and procedure tolerability in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Suspected prostate cancer eligible for transperineal prostate biopsy
* Patients who have signed informed consent
* Age > 50 years
* Male

Exclusion Criteria:

* patients who have had prostate biopsies in the past

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patients who need a prostate biopsy
Enrollment: 78 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
VAS pain scale | from start to the end of the procedure
  VAS pain scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang YH, Oh TH, Lee JW, Park SC, Seo IY, Jeong HJ, Kwon WA. Listening to music during transrectal ultrasound-guided prostate biopsy decreases anxiety, pain and dissatisfaction in patients: a pilot randomized controlled trial. Urol Int. 2015;94(3):337-41. doi: 10.1159/000368420. Epub 2014 Dec 18. PMID 25531837
- [Background] Dell'Atti L. Impact of music on anxiety and pain perception among men undergoing prostate biopsy: Synthesis of qualitative literature. Complement Ther Clin Pract. 2021 May;43:101330. doi: 10.1016/j.ctcp.2021.101330. Epub 2021 Feb 6. PMID 33578321
- [Background] Kyriakides R, Jones P, Geraghty R, Skolarikos A, Liatsikos E, Traxer O, Pietropaolo A, Somani BK. Effect of Music on Outpatient Urological Procedures: A Systematic Review and Meta-Analysis from the European Association of Urology Section of Uro-Technology. J Urol. 2018 May;199(5):1319-1327. doi: 10.1016/j.juro.2017.11.117. Epub 2017 Dec 7. PMID 29225059
- [Background] Vanoli S, Grobet-Jeandin E, Windisch O, Valerio M, Benamran D. Evolution of anxiety management in prostate biopsy under local anesthesia: a narrative review. World J Urol. 2024 Jan 20;42(1):43. doi: 10.1007/s00345-023-04723-2. PMID 38244150
- [Background] Novella G, Ficarra V, Galfano A, Ballario R, Novara G, Cavalleri S, Artibani W. Pain assessment after original transperineal prostate biopsy using a coaxial needle. Urology. 2003 Oct;62(4):689-92. doi: 10.1016/s0090-4295(03)00483-7. PMID 14550444